CLINICAL TRIAL: NCT05168943
Title: Nylon Versus Polyurethane Epidural Catheters In Patients Undergoing Major Orthopedic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour Teaching Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DTH: 21003
Record Dates: First submitted 2021-12-10; First posted 2021-12-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-06

CONDITIONS: Epidural; Anesthesia; Catheter Complications; Catheter Blockage; Catheter Dysfunction; Catheter Breakage
Keywords: Epidural Anesthesia; Nylon (Polyamide) Epidural Catheter; Polyurethane Epidural Catheter

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group N (n=30) (Active Comparator): Continuous Epidural Anesthesia using Nylon (Polyamide) Epidural Catheter
  Interventions: Device: Nylon (Polyamide) Epidural Catheter
- Group P (n=30) (Active Comparator): Continuous Epidural Anesthesia using Polyurethane Epidural Catheter
  Interventions: Device: Polyurethane Epidural Catheter

INTERVENTIONS:
Device: Nylon (Polyamide) Epidural Catheter — Nylon (Polyamide) Epidural Catheter
  Arms: Group N (n=30)
Device: Polyurethane Epidural Catheter — Polyurethane Epidural Catheter
  Arms: Group P (n=30)

SUMMARY:
Objectives: To compare the safety and efficacy of nylon (polyamide) epidural catheter versus polyurethane epidural catheter in patients undergoing major orthopedic surgery under continuous epidural anesthesia.

Background: Continuous epidural anesthesia is the most common anesthetic technique used in orthopedic surgery. However, the use of epidural catheters is associated with complications. The insertion of the catheter may be associated with intravascular or intrathecal placement, nerve root irritation, paresthesia, kinking, hematoma, or breakage during catheter removal.

Patients and Methods: This was a prospective, randomized, double-blind clinical trial; carried out on 60 patients undergoing major orthopedic surgery under continuous epidural anesthesia. Patients were randomly allocated into two equal groups; group N, using Nylon catheter, and group P, using Polyurethane catheter.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status ≤ II
* Age from 21 to 60 years
* Body Mass Index (BMI) < 35

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status > II
* Age < 21 years or > 60 years
* Body Mass Index (BMI) ≥ 35
* Contraindications to regional anesthesia (including coagulopathy and infection at the injection site)
* Uncooperative patients
* Patients with known allergy to local anesthetics or opioids

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean and Standard deviation of Time required for epidural catheter insertion (seconds) (mean±SD) | 2 minutes after identifying the epidural space by loss of resistance technique
  Time interval from holding the epidural catheter by the anesthetist till removal of the Tuohy needle through the epidural catheter by the anesthetist

SECONDARY OUTCOMES:
Mean and Standard deviation of Time required for epidural catheter to anchor with the catheter connector (seconds) (mean±SD) | 2 minutes after removal of the Tuohy needle through the epidural catheter
  Time interval from holding the epidural catheter by the anesthetist till anchoring it with the catheter connector by the anesthetist
Mean and Standard deviation of Time required for epidural catheter removal (seconds) (mean±SD) | 2 minutes after the end of the operation
  Time interval from holding the epidural catheter by the anesthetist till removal of the epidural catheter by the anesthetist
Number of participants and Rate of Catheter-related complications | 2 minutes after the end of the operation
  Number of participants and Rate of: Catheter kink, Catheter stretch, Difficult catheter insertion, Intravascular placement, Intrathecal placement, Paresthesia, Failure (asymmetric, unilateral, no block at 30 min), Hematoma, Breakage during removal.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Shaat, MD, Principal Investigator — Damanhour Teaching Hospital
Locations (1):
- Damanhour Teaching Hospital, Damanhūr, El-Beheira, Egypt